CLINICAL TRIAL: NCT02303756
Title: Colonic Capsule Endoscopy (CCE) for Screening of Neoplasm's
Brief Title: Colonic Capsule Endoscopy (CCE) for Screening of Neoplasm's A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Niels Qvist, Professor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20140141
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Rectal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pillcam® COLON Capsule (Experimental): Detection of neoplastic lesions in colon and rectum compared to colonoscopy
  Interventions: Device: Pillcam® COLON Capsule

INTERVENTIONS:
Device: Pillcam® COLON Capsule — colonoscopy

SUMMARY:
The primary aim is to evaluate the efficiency of capsule endoscopy (CCE) in in the detection of neoplasms compared to conventional colonoscopy in persons participating in the Danish screening program for colorectal cancer with a positive fecal occult blood with the colonoscopy being the gold standard.

DETAILED DESCRIPTION:
Participants will be recruited from the screening program, and are living on the main island of Funen. Persons with a positive FOBT who have been offered and have accepted a colonoscopy will be contacted by telephone and informed about the project by the project nurse.

The persons who accept participation and meet the inclusion criteria will be contacted by the study nurse for scheduling the capsule endoscopy according to the planned colonoscopy, which has to bee within 9-13 days after the result of the FOBT test.

The nurse will instruct the person to take the standard colon preparation 2 days before the colonoscopy, and stay from solid food until after the colonoscopy has been performed according to standard procedure. Thus the period with food-restrictions has to be extended by one day. A visit by the home services nurse the day before the colonoscopy will be arranged. The nurse will assist and supervise the intake of the video capsule and assists with the attachment of the monitor in a belt around the person's belly. Afterwards the questionnaire 1 (appendix 1) will be fulfilled by the patient with assistance from the nurse.

When the capsule has passed anus the monitoring equipment must be disarmed by the patient and stored according to the instructions. The patient will bring the recorder to the hospital the following day and deliver it to the study nurse, who will take care of data-transmission to the institute in Hamburg. After the colonoscopy and recovery period, the patient and the project nurse will fulfill the 2. questionnaire (appendix 2) and the colonoscopist will fulfill a standard report on the findings and treatment at colonoscopy (appendix 3), which will be added to the electronic database by the project secretary. The results form the colonoscopy will be the only information, that will be retrieved form the patients record.

Trained specialists in the Diagnostic Centre in Hamburg will perform the evaluation of the CCE and the data will be entered in a standard diagnostic report (appendix 4). The Diagnostic Centre will not have access to the results of the colonoscopy.

The CCE report must be available within 3 days, and the project responsible will evaluate the result according to the reported findings at colonoscopy. Any disagreement will be evaluated and discussed with the patient. In case of significant disagreement defined as a neoplasms of > 9 mm found at CCE and not detected by colonoscopy the patient will be offered additional diagnostics in the form of repeated colonoscopy within 2 weeks or a CT colonography upon the decision by the patient.

Participants have to stay on a fluid diet for one day more than for the conventional investigation. This might be uncomfortable for some patients, but is without any health-related risk. Another side effect could be increased fecal content in the bowel at colonoscopy due to the extended time from bowel preparation to colonoscopy. In some cases this could result in an incomplete colonscopy, which then has to be repeated. The risk of this side effect is unknown but is considered to be below 5%.

The most significant complication to the CCE will be the risk of impaction of the capsule within the intestine, which may lead to surgery. The risk is minimized by the exclusion criteria and according to daily clinical experience the risk will be less than 0.5%, and will mainly occur in persons with an unknown intestinal pathology, which in the majority of the cases would necessitate surgical treatment anyway. There is no known risk with the monitoring equipment.

In the case of significant disagreement between the results form capsule endoscopy and the conventional colonoscopy the patient may risk further investigations, but on the other hand this could be an advantage for the patients in case of missed lesions at the colonoscopy. The risk of missing cancer or large polyps by colonoscopy is in the range of 1-2%.

ELIGIBILITY:
Inclusion Criteria:

* Positive feaecal occult bleeding test at screening

Exclusion Criteria:

* Previous gastrointestinal surgery except for appendectomy
* Known inflammatory bowel disease including Chrohn's disease and ulcerative colitis
* An ostomy
* Symptoms on bowel obstruction (recurrent abdominal pain, constipation or vomiting within the last 3 months)
* Vomiting in connection with the bowel emptying procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Identification of neoplasia | One week after examination
  Compared to colonoscopy

SECONDARY OUTCOMES:
Completion rate | 24 hours
  Documented capsule excretion on the viedorecordin

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odesne University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Buijs MM, Kroijer R, Kobaek-Larsen M, Spada C, Fernandez-Urien I, Steele RJ, Baatrup G. Intra and inter-observer agreement on polyp detection in colon capsule endoscopy evaluations. United European Gastroenterol J. 2018 Dec;6(10):1563-1568. doi: 10.1177/2050640618798182. Epub 2018 Sep 11. PMID 30574327
- [Derived] Buijs MM, Kobaek-Larsen M, Kaalby L, Baatrup G. Can coffee or chewing gum decrease transit times in Colon capsule endoscopy? A randomized controlled trial. BMC Gastroenterol. 2018 Jun 25;18(1):95. doi: 10.1186/s12876-018-0824-9. PMID 29940864
- [Derived] Blanes-Vidal V, Nadimi ES, Buijs MM, Baatrup G. Capsule endoscopy vs. colonoscopy vs. histopathology in colorectal cancer screening: matched analyses of polyp size, morphology, and location estimates. Int J Colorectal Dis. 2018 Sep;33(9):1309-1312. doi: 10.1007/s00384-018-3064-0. Epub 2018 May 1. PMID 29717351